CLINICAL TRIAL: NCT00517543
Title: A Randomized, Open Label, 4 Period Crossover Study in Healthy Subjects to Determine the Effect of Particle Size on the Pharmacokinetics of a Single mg Dose of GW856553
Brief Title: A Study to Examine the Effect of Particle Size on Bioequivalence and Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 109385
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Rheumatoid Arthritis; Atherosclerosis
Keywords: inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Arthritis, Rheumatoid; Atherosclerosis; Inflammation | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

INTERVENTIONS:
Drug: GW856553

SUMMARY:
This study is being conducted to measure the amount of study drug that is in your blood after you receive a different type of tablet in each of four study visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females between 18 and 60 years of age, inclusive. Whether a subject is "healthy" will be determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring.
* To be eligible, female subjects must have a negative pregnancy test (i.e. serum hCG test) and be of:

  1. non-childbearing potential (i.e. physiologically incapable of becoming pregnant). This includes pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy, or documented hysterectomy - tubal ligation is not sufficient.
  2. childbearing potential and agrees to commit to two of the protocol-approved methods of contraception, when used consistently and in accordance with both the product label and the instructions of a physician (and as listed in Appendix 3).
* Male subjects must agree to abstain from or use a condom during sexual intercourse with pregnant or lactating females; or use a condom/spermicide, in addition to having their female partner use another form of contraception, such as an IUD, diaphragm with spermicide, oral contraceptive, inject able progesterone, or sub dermal implant if engaging in sexual intercourse with a female partner who could become pregnant. This criterion must be followed from the time of the first dose of study medication until completion of follow up procedures.
* Body weight >/ 50 kg (110 pounds) for men and >/ 45 kg (99 pounds) for women and body mass index (BMI) between 19 and 31.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and bilirubin within reference range at screening.
* Signed and dated written informed consent prior to admission to the study. The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination, or ECG (12 lead) judged by the Investigator and /or GSK medical monitor to potentially introduce additional risk factors and/or interfere with the study procedures.
* Significant cardiac, pulmonary, metabolic, renal, hepatic, neurological, psychiatric, or gastrointestinal conditions that in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as participant in this trial.
* History of Gilbert's syndrome.
* Elevated blood pressure or history of elevated blood pressure considered clinically significant by the Investigator.
* History of increased liver function tests [alanine aminotransferase (ALT), aspartate aminotransferase (AST) above 1.5 x upper limit of normal (UNL) in the past 6 months.
* History of alcohol/drug abuse or dependence within 12 months of the study.
* The subject has a positive pre-study drug or alcohol screen.
* Positive for Hepatitis C antibody, Hepatitis B surface antigen or HIV.
* History of regular alcohol consumption averaging > 7 drinks/week for women or > 14 drinks/week for men. One drink is equivalent to (12 g alcohol) = 5 ounces (150 mL) of wine; or 12 ounces (360 mL) of beer; or 1.5 ounces (45 mL) of 80 proof distilled spirits within 6 months of screening.
* Urinary cotinine levels indicative of smoking. History or regular use of tobacco or nicotine-containing products within 6 months prior to screening.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John'sWort, kava, ephedra (ma huang), gingko biloba, DHEA, yohimbe, saw palmetto, ginseng and red yeast rice) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Where participation in this study would result in donation of blood in excess of 500 mL within a 56-day period.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to dosing.
* Female subjects who are nursing, pregnant, or plan to become pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
1) to demonstrate bioequivalence of four different particle sizes by assay of blood from dosing through 72 hours post dose in each of four study periods

SECONDARY OUTCOMES:
1) determine/compare relative bioavailability by assay of blood (dosing to 72 hr in 4 study periods) 2) assess safety/tolerability of single oral doses thru AE reporting; vs & ECG monitoring from per 1 dosing thru study f/u
determine the relative bioavailability of a single oral dose of 15 mg GW856553 in healthy subjects using a tablet with a particle size of > 20 microns (a milled formulation) compared to tablets with particle sizes of 2 microns, 4 microns, and 6 microns.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States